CLINICAL TRIAL: NCT02089659
Title: A 2-Part, Open-Label, Singe-Dose Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of MK-1439
Brief Title: A Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of Doravirine (MK-1439) (MK-1439-019)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1439-019; MK-1439-019 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-07

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Moderate Hepatic Insufficiency (Experimental): Participants with moderate hepatic insufficiency receive a single oral dose of 100 mg doravirine on Day 1 of Part 1. All participants in this arm were to have moderate hepatic insufficiency based on the Child-Pugh scale.
  Interventions: Drug: Doravirine
- Part 1: Healthy Matched Control (Experimental): Healthy participants matched for age and weight receive a single oral dose of 100 mg doravirine on Day 1 of Part 1.
  Interventions: Drug: Doravirine
- Part 2: Mild Hepatic Insufficiency (Experimental): Participants with mild hepatic insufficiency receive a single oral dose of 100 mg doravirine on Day 1 of Part 1. All participants in this arm were to have mild hepatic insufficiency based on the Child-Pugh scale. This arm was to be enrolled and investigated only if a clinically meaningful increase in exposure of doravirine was observed in participants with moderate hepatic insufficiency in Part 1.
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — Following an overnight fast, a single tablet of 100 mg doravirine was be administered orally
  Other Names: MK-1439

SUMMARY:
This study aimed to investigate the influence of hepatic insufficiency on the pharmacokinetics (PK) of doravirine (MK-1439). In Part 1, PK of doravirine in participants with moderate hepatic insufficiency was compared with that of healthy control subjects matched with regard to mean age and weight. If a clinically meaningful increase in exposure of doravirine was observed in participants with moderate hepatic insufficiency in Part 1, study Part 2 was to evaluate PK of doravirine in participants with mild hepatic insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 19 and 40 kg/m^2
* Continuous non-smoker or moderate smoker of <20 cigarettes or equivalent per day. Agrees to consume <=10 cigarettes or equivalent per day from the time of screening through the period of sample collection.
* In good health and with no clinically significant electrocardiogram abnormality
* Hepatic impairment participants: diagnosis of chronic (>6 months), stable hepatic insufficiency with features of cirrhosis due to any etiology. Part 1 only: score of 7 to 9 on the Child-Pugh scale. Part 2: score of 5 to 6 on the Child-Pugh scale.
* Females of childbearing potential: sexually inactive for >=14 days before study drug administration and throughout the study, or using 2 acceptable methods of barrier contraception from screening until 14 days after study drug administration.

Exclusion Criteria:

* Mentally or legally incapacitated or has significant emotional problems at the time of screening or expected during the study
* History or presence of clinically significant medical or psychiatric condition or disease
* History or presence of drug abuse within the past 2 years
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds
* Female participant who is pregnant or lactating
* Positive results for breath alcohol or urine drug screen (unless due to prescription drug use and is approved by the investigator) at screening
* Positive for HIV at screening
* Unable to refrain from or anticipates the use of any drug known to be a significant inhibitor or inducer of cytochrome oxidase CYP3A or P-glycoprotein, or any medication or substance which cannot be discontinued at least 14 days before study drug administration and throughout the study.
* Donation of >500 mL of blood or had significant blood loss within 56 days before study drug administration
* Plasma donation within 7 days before study drug administration
* Dosed in another clinical trial within 28 days before study drug administration
* Healthy control participants only: positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) at screening;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2014-05-12 (Actual); Study Completion 2014-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinicaltrials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Khalilieh S, Yee KL, Liu R, Fan L, Sanchez RI, Auger P, Triantafyllou I, Stypinski D, Lasseter KC, Marbury T, Iwamoto M. Moderate Hepatic Impairment Does Not Affect Doravirine Pharmacokinetics. J Clin Pharmacol. 2017 Jun;57(6):777-783. doi: 10.1002/jcph.857. Epub 2016 Dec 27. PMID 28026013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 2 of the study was to enroll participants only if a clinically meaningful increase in exposure of doravirine was observed in participants with moderate hepatic insufficiency in Part 1. Because this was not observed, no participants were enrolled in Part 2 of the study.
Groups:
- Part 1: Participants With Moderate Hepatic Insufficiency: Participants with moderate hepatic insufficiency received a single oral dose of 100 mg doravirine on Day 1 of Part 1. All participants in this arm were to have moderate hepatic insufficiency based on the Child-Pugh scale.
- Part 1: Healthy Control Participants: Healthy participants matched for age and weight received a single oral dose of 100 mg doravirine on Day 1 of Part 1.
- Part 2: Participants With Mild Hepatic Insufficiency: Participants with mild hepatic insufficiency received a single oral dose of 100 mg doravirine on Day 1 of Part 1. All participants in this arm were to have mild hepatic insufficiency based on the Child-Pugh scale. This arm was to be enrolled and investigated only if a clinically meaningful increase in exposure of doravirine was observed in participants with moderate hepatic insufficiency in Part 1.
Period: Overall Study
Arm/Group | Part 1: Participants With Moderate Hepatic Insufficiency | Part 1: Healthy Control Participants | Part 2: Participants With Mild Hepatic Insufficiency
Started | 8 | 8 | 0
Completed | 8 | 8 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Participants With Moderate Hepatic Insufficiency | Part 1: Healthy Control Participants | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: Years] | 59 [54 to 64] | 56 [44 to 63] | 57 [44 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12
Child-Pugh Total Score [Count of Participants; unit: Participants] — The Child-Pugh scale was used to classify the severity of liver disease in study participants. The total score is the sum of the scores on 5 clinical measures of liver disease, each on a 3-point scale where 3 is greatest severity: total bilirubin, serum albumin, INR, ascites, and hepatic encephalopathy. The total Child-Pugh score ranges from 5 to 15, where a score of 7 to 9 represents moderate hepatic insufficiency. Population: All enrolled participants. Healthy participants were not evaluated for Child-Pugh scores.
  Participants
    number analyzed (Participants) | 8 | 0 | 8
    Total Score = 7 | 2 | 0 | 2
    Total Score = 8 | 4 | 0 | 4
    Total Score = 9 | 2 | 0 | 2
Weight [Mean (Full Range); unit: kg] | 82.0 [55.6 to 119.0] | 79.8 [66.0 to 92.1] | 80.9 [55.6 to 119.0]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 Hours to Infinity (AUC0-∞) of Doravirine
Description: Blood was collected for the determination of plasma doravirine using a liquid chromatographic tandem mass spectrometric method
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 6, 12, 24, 48, and 72 hours postdose for all participants and at 96, 120, and 144 hours postdose for participants with hepatic insufficiency
Population: The analysis population consisted of the subset of participants who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part 1: Participants With Moderate Hepatic Insufficiency | Part 1: Healthy Control Participants
Number analyzed (Participants) | 8 | 8
µM*hr | 53.9 [41.5 to 70.0] | 54.6 [42.1 to 71.0]
Statistical Analysis 1: Comparison: Part 1: Participants With Moderate Hepatic Insufficiency vs Part 1: Healthy Control Participants; Test type: Other; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.72 to 1.35] — Moderate hepatic insufficiency / Healthy controls

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Doravirine
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Part 1: Participants With Moderate Hepatic Insufficiency | Part 1: Healthy Control Participants
Number analyzed (Participants) | 8 | 8
nM | 1850 [1420 to 2420] | 2050 [1570 to 2680]
Statistical Analysis 1: Comparison: Part 1: Participants With Moderate Hepatic Insufficiency vs Part 1: Healthy Control Participants; Test type: Other; Geometric Mean Ratio = 0.90, 90% CI 2-sided [0.66 to 1.24] — Moderate hepatic insufficiency / Healthy controls

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Form 0 to 24 Hours (AUC0-24) of Doravirine
Description: as for outcome 1
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 6, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part 1: Participants With Moderate Hepatic Insufficiency | Part 1: Healthy Control Participants
Number analyzed (Participants) | 8 | 8
µM*hr | 28.5 [23.4 to 34.8] | 30.6 [25.1 to 37.3]
Statistical Analysis 1: Comparison: Part 1: Participants With Moderate Hepatic Insufficiency vs Part 1: Healthy Control Participants; Test type: Other; Geometric Mean Ratio = 0.93, 90% CI 2-sided [0.74 to 1.18] — Moderate hepatic insufficiency / Healthy controls

4. Primary Outcome: Plasma Concentration of Doravirine at 24 Hours (C24)
Description: as for outcome 1
Time Frame: 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Part 1: Participants With Moderate Hepatic Insufficiency | Part 1: Healthy Control Participants
Number analyzed (Participants) | 8 | 8
nM | 842 [658 to 1080] | 847 [662 to 1080]
Statistical Analysis 1: Comparison: Part 1: Participants With Moderate Hepatic Insufficiency vs Part 1: Healthy Control Participants; Test type: Other; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.74 to 1.33] — Moderate hepatic insufficiency / Healthy controls

ADVERSE EVENTS:
Time Frame: Up to 14 days after drug administration
Description: The population analyzed was all participants who received at least 1 dose of study treatment.
Arm/Group | Part 1: Participants With Moderate Hepatic Insufficiency | Part 1: Healthy Control Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Participants With Moderate Hepatic Insufficiency (N=8) | Part 1: Healthy Control Participants (N=8)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.